CLINICAL TRIAL: NCT04772391
Title: Fitness Intervention Trial in Adults With Sickle Cell Disease (SCD Fit): A Feasibility Study
Brief Title: Fitness Trial in Adults With Sickle Cell Disease (SCD Fit): A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300006888
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Cardiovascular Diseases; Sickle Cell Disease; Exercise
MeSH Terms: conditions — Cardiovascular Diseases; Anemia, Sickle Cell; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Treatment Group (Other): Exercise Sessions
  Interventions: Other: Exercise Sessions

INTERVENTIONS:
Other: Exercise Sessions — Participant will complete up to 8 exercise sessions

SUMMARY:
The purpose of this project is to develop novel approaches to promote health and longevity while enhancing quality of life among persons with Sickle cell disease (SCD). Therefore, investigators are aiming to adapt an evidence-based exercise intervention for adults with SCD informed by culturally- relevant and biologic factors and pre-test the adapted exercise program in a small sample of adults with SCD.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a major public health concern as it is the most common inherited blood disorder in the US, affecting over 100,000 persons.(1) This disease predominantly affects African Americans, occurring in 1 out 365 African American births. Sickle cell disease causes intermittent extremely painful vaso-occlusion events, which lead to multi-organ damage, significant morbidity and early mortality - and resulting in increased healthcare utilization with estimated annual United States healthcare costs of 786 million.(2,3) To date, there are very few strategies for reducing pain, preventing organ dysfunction, and improving quality of life for persons with SCD leading to a disproportionate disparity in care. For this reason, there is a critical need to develop novel approaches to promote health and longevity while enhancing quality of life among persons with SCD.

Exercise capacity and cardiorespiratory fitness are important predictors of cardiovascular outcomes and overall survival; however, adults with SCD have severely reduced levels of fitness, with less than 50% of expected compared to the general population. (4) Since cardiopulmonary disease accounts for 40% of the mortality in adults with SCD, enhancing physical activity with regular exercise is one potential method for improving survival, reducing poor Cardiovascular disease (CVD) outcomes, and improving quality of life for adults with SCD.(5,6) Evidence-based exercise interventions in rheumatoid arthritis, an inflammatory, chronic disease with similar sequelae to SCD, have shown that exercise interventions can increase quality of life, reduce pain, and improve CVD outcomes.(7-9) Currently, a paucity of research on the benefits of exercise for SCD exists and this is a critical barrier to overcome to both understand the role of physical fitness SCD and to develop evidence-based recommendations to guide exercise in SCD. Only one small study of an exercise intervention program in France has reported exercise to be safe, effective, and reverse SCD-related muscle vasculature damage but long term data in larger populations are needed.(10) Therefore, there is a need to conduct more studies in the United States and to develop an evidence-based exercise program for adults with SCD that integrates patient perspectives, can be broadly implemented among different settings, and is physically safe. To address this unmet need, the central hypothesis of this proposal is that an evidence-based exercise intervention informed by the needs and preferences of adults with SCD will be feasible, acceptable, and tolerable in a cohort of adults with SCD. Our long-term goal is to develop a safe and effective exercise intervention to promote sustainable physical activity in SCD and to guide exercise recommendations for SCD which currently do not exist. Therefore, investigators propose to adapt an evidence-based exercise intervention for adults with SCD informed by culturally- relevant and biologic factors and pre-test the adapted exercise program in a small sample of adults with SCD.

Outcomes: The primary outcome will be to collect preliminary data on feasibility, acceptability, and tolerability of the exercise intervention. Rates of recruitment and retention will be measured to assess feasibility. Acceptability will be measured through attendance, engagement, and qualitative feedback. Tolerability will be measured by the ability for participants to complete the exercise program without adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have sickle cell disease of any genotype
* Participant must be 18 years of age
* Participant must be seen and followed by the UAB sickle cell center
* Participant must have reliable transportation to the UAB center of Exercise Medicine
* Participant must be in steady-state disease (No vaso-occlusive crisis or SCD-related hospitalization with 4 weeks of enrollment)

Exclusion Criteria:

* Participant has avascular necrosis
* Participant is pregnant
* Participant has absolute contraindications to exercise according to the American Heart Association and American College of Sports Medicine guidelines (42)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Feasibility will be measured | One year
  Outcome will be to collect preliminary data on feasibility of the exercise intervention using rates of recruitment and retention
Acceptability will be measured | One year
  Outcome will be to collect preliminary data on acceptability of the exercise intervention using attendance, engagement, and qualitative feedback.
Tolerability will be measured | One year
  Outcome will be to collect preliminary data on tolerability of the exercise intervention using the ability for participants to complete the exercise program without adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Foluso Ogunsile, MD, Principal Investigator — Memorial Healthcare System
Locations (1):
- Memorial Healthcare System, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No
To be determined